CLINICAL TRIAL: NCT00352599
Title: Trial to Evaluate the Safety of Lovastatin in Individuals With Neurofibromatosis Type I (NF1)
Acronym: NF1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05-08-069-01
Record Dates: First submitted 2006-07-13; First posted 2006-07-14 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Neurofibromatosis 1
Keywords: Neurofibromatosis Type 1; NF1; Lovastatin; statin
MeSH Terms: conditions — Neurofibromatosis 1 | interventions — Lovastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lovastatin (Active Comparator): Lovastatin
  Interventions: Drug: Lovastatin
- Placebo pill (Placebo Comparator): Placebo pill
  Interventions: Drug: placebo pill

INTERVENTIONS:
Drug: Lovastatin
  Arms: Lovastatin
Drug: Lovastatin — Lovastatin capsules daily for 14 weeks (titrated up from 10 mg to 40 mg)
  Arms: Lovastatin
Drug: placebo pill
  Arms: Placebo pill

SUMMARY:
Neurofibromatosis type I (NF1) is a genetic disorder that affects approximately 1 in 3500 individuals. Half of people with NF1 inherit the condition from a parent, and half have a new occurrence of the condition. The manifestation of NF1 is highly variable and multiple organ systems are typically affected. Some of the more common symptoms include benign neurofibromas, café au lait spots, Lisch nodules (tan spots on the iris of the eye). Some individuals with NF1 also exhibit more severe associated conditions, such as optic pathway tumors (gliomas) or bones bending or curving. Neurocognitive deficits and specific learning disabilities occur in approximately 30 to 50% of individuals with NF1 and are regarded by some observers and sufferers to be among the most troubling features of a disease. The most commonly reported findings are deficits in visuoperceptual ability, motor coordination, expressive and receptive language, and executive functioning, which requires intact short-term memory and attention. Patients with NF1 also show a slight depression in mean IQ scores compared to healthy adults without the disorder.

While cognitive deficits are now a widely-recognized feature of Neurofibromatosis Type 1 (NF1), the precise cause of these deficits still remain to be determined. Dr. Alcino Silva, a co- investigator on this study, has developed an animal model of NF1 in which mice have a specific mutation of the *NF1* gene. These mice are physically normal but show specific learning impairments. Dr. Silva's lab found that treatment with a medication called lovastatin, a drug typically used for high cholesterol, reversed some of the spatial deficits seen in these animals. Lovastatin is a medication commonly used to treat high cholesterol and has been proven to be relatively safe and tolerable in humans.

The investigators are now conducting a randomized, double-blinded, placebo- controlled, trial of lovastatin in patients with NF1. Participants will be randomly assigned to lovastatin or placebo and treated for approximately 14 weeks with baseline and follow-up assessments to evaluate safety and any effects on neurocognitive test performance.

ELIGIBILITY:
Inclusion Criteria:

1. a diagnosis of NF1 by NIH criteria
2. between 10 and 50 years of age
3. no evidence of a comorbid neurological disorder (e.g., epilepsy, encephalitis)
4. not currently taking a statin medication
5. not suffering from hypercholesterolemia based on self-report, collateral information from physician, or initial medical workup using National Cholesterol Education Program (NCEP, JAMA 2001), guidelines accepted by the American College of Cardiology (ACC) and the American Heart Association (AHA)
6. does not have any of the aforementioned conditions that contraindicates use of statin medications (such as pregnancy, lactation, liver disease, or use of other medication not recommended for use in conjunction with lovastatin). A negative pregnancy test will be required if the patient is a female in reproductive years.
7. not mentally retardation (i.e., IQ greater than 70)
8. no evidence of significant and habitual alcohol or drug abuse or dependence
9. sufficient acculturation and fluency in the English language to avoid invalidating research measures of thought, language, and speech disorder, and verbal abilities.
10. lives in Southern California area (or can arrange ~5 visits to Los Angeles over 14 weeks)

Exclusion Criteria:

1. comorbid neurological conditions
2. significant drug or alcohol abuse
3. non-fluency in English

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2009-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Non-verbal learning /working memory | 14 weeks

SECONDARY OUTCOMES:
attention | 14 weeks
tolerability of medication | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carrie E Bearden, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Semel Institute for Neuroscience and Human Behavior, Los Angeles, California, United States

REFERENCES:
- [Background] Li W, Cui Y, Kushner SA, Brown RA, Jentsch JD, Frankland PW, Cannon TD, Silva AJ. The HMG-CoA reductase inhibitor lovastatin reverses the learning and attention deficits in a mouse model of neurofibromatosis type 1. Curr Biol. 2005 Nov 8;15(21):1961-7. doi: 10.1016/j.cub.2005.09.043. PMID 16271875
- [Background] Shilyansky C, Karlsgodt KH, Cummings DM, Sidiropoulou K, Hardt M, James AS, Ehninger D, Bearden CE, Poirazi P, Jentsch JD, Cannon TD, Levine MS, Silva AJ. Neurofibromin regulates corticostriatal inhibitory networks during working memory performance. Proc Natl Acad Sci U S A. 2010 Jul 20;107(29):13141-6. doi: 10.1073/pnas.1004829107. Epub 2010 Jul 12. PMID 20624961